CLINICAL TRIAL: NCT04646980
Title: Dietary Supplementation With Biobran/MGN-3 Increases Innate Resistance Against Viral Infections That Cause Influenza-like Illnesses in Elderly Subjects: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Biobran/MGN-3 Increases Innate Resistance and Reduces the Incidence of Influenza-like Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: Charles Drew University of Medicine and Science (Other); University of California, Irvine (Other); Daiwa Pharmaceutical Corporation Co, Ltd, Tokyo 154-0024 Japan (Unknown)
Responsible Party: Principal Investigator, Ahmed Farouk Elsaid, Assistant Professor of Community Medicine and Public Health, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4034-12-6-2018
Record Dates: First submitted 2020-11-15; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Influenza-like Illness
Keywords: Biobran/MGN-3; Old adults; influenza-like illness; NK cells activity; Degranulation assay; RIG-1, MDA5, ISG15, MX1
MeSH Terms: conditions — gaze palsy, familial horizontal, with progressive scoliosis; Diabetes Mellitus, Insulin-Dependent, 19 | interventions — polysaccharide MGN3

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biobran/MGN-3 (Experimental): This arm consisted from 20 males and 20 females. Biobran/MGN-3 was orally supplemented at dose of 500 mg per day for 3 months (end of November 2018- end of February 2019).
  Interventions: Dietary Supplement: Biobran/MGN-3
- Placebo (Placebo Comparator): This arm consisted from 20 males and 20 females. Placebo, with the same appearance and taste, was orally supplemented at dose of 500 mg per day for 3 months (end of November 2018- end of February 2019).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Biobran/MGN-3 — Biobran/MGN3 is defined by the Medicines and Healthcare products Regulatory Agency (MHRA) as a food supplement. Biobran/MGN3 is manufactured by hydrolyzing rice bran with the enzymatic extract of medicinal Shiitake mushrooms. Enzyme hydrolysis of rice bran produces arabinoxylane, a hemi-cellulose compound, which constitutes the active ingredient of biobran/MGN3.
  Arms: Biobran/MGN-3
Other: Placebo — Placebo, with same appearance and taste as Biobran/MGN-3, was given to control subjects at a dose of 500 mg everyday for 3 months
  Arms: Placebo

SUMMARY:
Influenza is a seasonally-epidemic viral infection causing 3-5 million severe illnesses and up to approximately 500,000 annual deaths around the world. Influenza-like illnesses (ILI) is a simple constellation of symptoms and signs that was introduced to capture influenza cases in surveillance system. The elderly are more susceptible to cancers and viral infections including influenza infection and complications that was attributed to the phenomenon of immunosenescence or age-associated decline of immune system activity. Biobran/MGN3 is a natural nutritional supplement that was shown to exhibit potent immunomodulator effect such as enhancement of natural killer cell (NKC) activity and up-regulating the production of cytokines such as tumor necrosis factor-α (TNF- α), interferon-gamma (IFN-γ) and -lambda (IFN-λ). The protective effect of Biobran/MGN-3 against viral infection such hepatitis C virus (HCV) and human immunodeficiency virus (HIV) as well as several cancer types has been previously reported in experimental animal models and humans. The objective of the current study was to investigate the effect of Biobran/MGN-3 on some innate immune system components and the incidence of ILI in the older adult population. The studied innate immune system included NKC activity and the expressions of intracellular viral nucleic acid sensors such as retinoic acid-inducible gene 1 (RIG-1), melanoma differentiation-associated protein 5 (MDA5) and some of their downstream signals such as ISG15 and MX1.

DETAILED DESCRIPTION:
The current study investigated the effect of oral supplementation with Biobran/MGN-3, 500 mg every day for 3 months, on several components of innate immune system and the incidence rate of influenza-like illnesses (ILI) in older adults population. The study protocol conformed to the ethical guidelines of the 1975 Declaration of Helsinki and was approval by Institutional Review Board (IRB) at the Faculty of Medicine, Zagazig University, Egypt. Zagazig University Hospitals serves over 1 million residents in Zagazig district and neighboring towns.

The study spanned the time period from November 2018 till the end of February 2019, a period with known peak incidence of ILI attacks. Subjects of ≥ 56 years were recruited from the visitors of outpatient clinics at Zagazig University Hospitals. The age of ≥ 56 years was used by the WHO to define old age in African nations. In addition, this age is close to public service retirement in Egyptian society, which is associated with significant social, mental, and psychological stress and therefore could be associated with significant decline in NK cell activity. Only local residents of Zagazig district were recruited to the study so as to reduce the dropout rate.

Originally 90 subjects, both males and females, were approached but only 80 subjects, 40 males and 40 females, continued the study. Ten of the recruits refused to participate when they realized that the sachets were only labeled with the manufacture symbols without printed names, which was used to ensure double-blinding. Informed consents were obtained from all participants and their right to unconditionally withdraw from the study at any time were made clear to them.

Males and females were randomly assigned into two groups (n=40/group) that received either placebo or Biobran/MGN-3 (500 mg/day for 3 months). Both the health care giver and the participants were blinded to the ingested supplement. Participants' health was monitored via weekly home visits and they were instructed to report any complaints or side effects by phone to the health care giver.

Diagnosis of ILI was made by documenting the incidence of acute respiratory illness with a measured temperature of ≥ 38 °C with cough (3). After diagnosis, the subject was helped to follow the proper health management plan by the health care giver. During the study, all participants were required not to take any vitamins or medications during the study without consultation.

The effect of Biobran/MGN-3 on liver, kidney, and hematological parameters were monitored. Liver functions were monitored using alanine aminotransferase (ALT/SGPT) and aspartate aminotransferase (AST/SGOT), whereas kidney function was monitored using serum uric acid. The assessed hematological parameters included red blood cell count (RBC), hematocrit value (HCT), hemoglobin (Hb), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), and total and differential (WBC).

NKC activity was measured using the well documented degranulation assay. The viral nucleic acid receptors, RIG-1 and MDA5, and their downstream target, ISG15 and MX1, were assessed using flowcytometry in BEAS-2B cells.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 56+ years
* Both sexes will be included.
* Local residents of Zagazig district
* Willing to participate in the study and give a written consent.

Exclusion Criteria:

* Subjects who took influenza vaccine, cortisone, or any other immunosuppressive agents such as radiation or chemotherapy.
* Diagnosed with infections or malignancies
* Presence of auto-immune disorders
* Marked portal hypertension, pancytopenia, renal, or kidney failure
* Presence of major psychological insult or under medication for psychological insult

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
ILI incidence rate | 12 weeks
  Incidence rate was calculated by dividing the number of incident ILI cases by the total number of the group participants during the 3 months study period.
ILI incidence density | 3600 Person-days
  incidence density was calculated by dividing the number of incident cases by the total person-time at risk
NK cell activity | 12 weeks
  Percentage of NK cells (CD56-positive CD3-negative) expressing CD-107a
RIG-1, MDA5, ISG15, MX1 expression | 72 hours
  Expression levels in BEAS-2B cells tissue culture exposed to Biobran/MGN-3

SECONDARY OUTCOMES:
Natural killer T-cells (NKT) cell activity | 12 weeks
  Percentage of NK cells (CD56-positive CD3-positive) expressing CD-107a

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Elsaid, MD/PhD, Principal Investigator — Department of Community Medicine and Public Health, Faculty of Medicine, Zagazig University
Locations (1):
- Department of Community Medicine and Public Health, Faculty of Medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Share results upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon request

REFERENCES:
- [Result] Elsaid AF, Shaheen M, Ghoneum M. Biobran/MGN-3, an arabinoxylan rice bran, enhances NK cell activity in geriatric subjects: A randomized, double-blind, placebo-controlled clinical trial. Exp Ther Med. 2018 Mar;15(3):2313-2320. doi: 10.3892/etm.2018.5713. Epub 2018 Jan 8. PMID 29456638
- [Result] Elsaid AF, Fahmi RM, Shaheen M, Ghoneum M. The enhancing effects of Biobran/MGN-3, an arabinoxylan rice bran, on healthy old adults' health-related quality of life: a randomized, double-blind, placebo-controlled clinical trial. Qual Life Res. 2020 Feb;29(2):357-367. doi: 10.1007/s11136-019-02286-7. Epub 2019 Sep 5. PMID 31489525

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04646980/Prot_SAP_000.pdf